CLINICAL TRIAL: NCT01123707
Title: A Multicenter, 52-week, Open-label Study to Assess the Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Patients With Major Depressive Disorder
Brief Title: To Assess the Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Participants With Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to Sponsor decision; no safety issues.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31-08-257; 2010-018860-17 (EudraCT Number)
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Aripiprazole; Escitalopram

STUDY DESIGN:
Intervention Model Description: Group composed of eligible rollover participants who completed one of the previous studies: 31-08-255 [NCT01111539], 31-08-256 [NCT01111552], or 31-08-263 [NCT01111565]
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Prior Aripiprazole/Escitalopram Combination Therapy (Experimental): Aripiprazole capsules, orally at the daily dose of 3, 6, or 12 mg, in combination with escitalopram 10 or 20 mg orally, once daily in combination with escitalopram 10 or 20 mg (i.e., the final dose taken during the previous study), orally, once daily, for 36 weeks. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 1 if the initial 6 mg/day dose was tolerated. The dose adjustments were allowed for aripiprazole to establish the maximum tolerated dose (MTD) by Week 4. Participants who received aripiprazole/escitalopram combination therapy in the double-blind treatment period in previous studies were included in this group.
  Interventions: Drug: Aripiprazole; Drug: Escitalopram
- Prior Escitalopram (Experimental): Aripiprazole capsules, orally at the daily dose of 3, 6, or 12 mg, in combination with escitalopram 10 or 20 mg orally, once daily in combination with escitalopram 10 or 20 mg (i.e., the final dose taken during the previous study), orally, once daily, for 36 weeks. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 1 if the initial 6 mg/day dose was tolerated. The dose adjustments were allowed for aripiprazole to establish the MTD by Week 4. Participants who received escitalopram in the double-blind treatment period in previous studies were included in this group.
  Interventions: Drug: Aripiprazole; Drug: Escitalopram
- Prior Aripiprazole (Experimental): Aripiprazole capsules, orally at the daily dose of 3, 6, or 12 mg, in combination with escitalopram 10 or 20 mg orally, once daily in combination with escitalopram 10 or 20 mg (i.e., the final dose taken during the previous study), orally, once daily, for 36 weeks. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 1 if the initial 6 mg/day dose was tolerated. The dose adjustments were allowed for aripiprazole to establish the MTD by Week 4. Participants who received aripiprazole in the double-blind treatment period in previous studies were included in this group.
  Interventions: Drug: Aripiprazole; Drug: Escitalopram
- Prior Single-blind Escitalopram (Experimental): Aripiprazole capsules, orally at the daily dose of 3, 6, or 12 mg, in combination with escitalopram 10 or 20 mg orally, once daily in combination with escitalopram 10 or 20 mg (i.e., the final dose taken during the previous study), orally, once daily, for 36 weeks. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 1 if the initial 6 mg/day dose was tolerated. The dose adjustments were allowed for aripiprazole to establish the MTD by Week 4. Participants who received escitalopram in the single-blind treatment period in previous studies were included in this group.
  Interventions: Drug: Aripiprazole; Drug: Escitalopram

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole oral capsules
  Other Names: OPC-14597
Drug: Escitalopram — Escitalopram oral capsules

SUMMARY:
This is a multicenter, 52-week, open-label study designed to assess the safety and tolerability of an oral aripiprazole/escitalopram combination therapy in outpatients with major depressive disorder (MDD). Enrollment into the study will be from eligible participants who have completed participation in Protocol 31-08-255 [NCT01111539], 31-08-256 [NCT01111552], or 31-08-263 [NCT01111565] ("rollover" participants).

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in Protocol 31-08-255, 31-08-256, or 31-08-263.

Exclusion Criteria:

* Participants with a current need for involuntary commitment or who have been hospitalized ≤ 28 days of the Baseline Visit for the current major depressive episode.
* Participants with a diagnosis of delirium, dementia, amnestic or other cognitive disorder, schizophrenia, schizoaffective disorder, or other psychotic disorder, Bipolar I or II disorder, eating disorder (including anorexia nervosa or bulimia), obsessive compulsive disorder, panic disorder, or posttraumatic stress disorder.
* Participants with a diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.
* Participants experiencing hallucinations, delusions, or any psychotic symptomatology in the current depressive episode.
* Participants who have met Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for substance abuse in the past 6 months (prior to the Baseline Visit) and/or dependence up to and including the past 12 months (prior to the Baseline Visit), including alcohol and benzodiazepines, but excluding caffeine and nicotine. Participants with two positive drug results for cocaine should be excluded from the study.
* Participants with hypothyroidism or hyperthyroidism.
* Participants with a significant risk of committing suicide based on history, investigator's judgment, and/or evaluation based on the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Participants who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders.
* Participants with insulin-dependent diabetes mellitus (IDDM).
* Participants with epilepsy or significant history of seizure disorders, except for a single childhood febrile seizure, post-traumatic, etc.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-11-18 (Actual); Primary Completion 2011-09-27 (Actual); Study Completion 2011-09-27 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 67 investigative sites in Australia, Estonia, India, Mexico, South Korea, and the United States from 18 November 2010 to 27 September 2011.
Pre-assignment Details: A total of 173 participants from studies 31-08-255 (NCT01111539), 31-08-256 (NCT01111552), and 31-08-263 (NCT01111565) were enrolled, of which 170 participants received aripiprazole/escitalopram combination therapy and were analyzed in this 31-08-257 study (NCT01123707). The data is reported as per the treatment received in previous studies.
Period: Overall Study
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Started | 44 | 41 | 38 | 50
Safety Sample (Participants who received at least one dose of aripiprazole/escitalopram combination therapy.) | 44 | 41 | 36 | 49
Completed | 0 | 0 | 0 | 0
Not Completed | 44 | 41 | 38 | 50
Not completed — Lost to Follow-up | 3 | 1 | 3 | 2
Not completed — Adverse Event | 5 | 7 | 5 | 3
Not completed — Sponsor Discontinued Study | 30 | 24 | 25 | 40
Not completed — Participant Met Withdrawal Criteria | 1 | 1 | 0 | 1
Not completed — Investigator Withdrew Participant | 0 | 1 | 1 | 1
Not completed — Subject Withdrew Consent | 4 | 5 | 1 | 2
Not completed — Lack of Efficacy | 1 | 2 | 1 | 0
Not completed — Subject Met Exclusion Criteria | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record.
Groups:
- Prior Aripiprazole/Escitalopram Combination Therapy: Aripiprazole capsules, orally at the daily dose of 3, 6, or 12 mg, in combination with escitalopram 10 or 20 mg orally, once daily in combination with escitalopram 10 or 20 mg (i.e., the final dose taken during the previous study), orally, once daily, for 36 weeks. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 1 if the initial 6 mg/day dose was tolerated. The dose adjustments were allowed for aripiprazole to establish the MTD by Week 4. Participants who received aripiprazole/escitalopram combination therapy in the double-blind treatment period in previous studies were included in this group.
- Total: Total of all reporting groups
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram | Total
Number analyzed (Participants) | 44 | 41 | 36 | 49 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (12.0) | 45.8 (10.7) | 48.6 (10.8) | 43.4 (11.3) | 45.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 25 | 26 | 33 | 118
  Male | 10 | 16 | 10 | 16 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 4 | 5 | 24
  Not Hispanic or Latino | 36 | 34 | 32 | 43 | 145
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 5 | 5 | 24
  White | 33 | 31 | 30 | 42 | 136
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (STEAEs), Severe (Grade 3 or Higher) TEAEs, and Discontinuations From the Trial Due to TEAEs
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it did not necessarily have to have a causal relationship with this treatment. An AE was considered serious if it was fatal; life-threatening; persistently or significantly disabling or incapacitating; required in-patient hospitalization or prolonged hospitalization; a congenital anomaly/birth defect; or other medically significant event that, based upon appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention. TEAE is defined as an adverse event that started after start of study drug treatment. The Common Terminology Criteria for Adverse Events v3.0 (CTCAE) was used to determine the severity wherein Grade 1=mild AE, Grade 2=moderate AE, Grade 3=severe AE, Grade 4=life-threatening or disabling AE, Grade 5=death related to AE.
Time Frame: From first dose up to 30 days post last dose (Up to approximately 40 weeks)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
percentage of participants
  TEAEs | 54.5 | 70.7 | 75.0 | 67.3
  STEAEs | 2.3 | 9.8 | 0.0 | 0.0
  Severe (Grade 3 or Higher) TEAEs | 0.0 | 4.9 | 5.6 | 2.0
  Discontinuations from the Trial due to TEAEs | 11.4 | 17.1 | 13.9 | 6.1

2. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression - Severity of Illness Scale (CGI-S) Score
Description: The severity of illness was rated using a 7-point CGI-S. CGI-S scores range from 1 to 7, where 1=normal, not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill participants. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 14, 20, 26, 32 and End of the study visit (Week 43 or before)
Population: Intent-to-treat (ITT) Sample included all participants in the Safety Sample with at least one CGI-S assessment in the Treatment Phase, with data available for analysis. Number analyzed is the number of participants with data available at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 48
score on a scale
  Baseline | 3.1 (1.1) | 3.4 (1.2) | 3.4 (0.9) | 3.2 (0.7)
  Change from Baseline at Week 1: number analyzed (Participants) | 42 | 40 | 33 | 45
  Change from Baseline at Week 1 | -0.0 (0.7) | -0.2 (0.6) | -0.2 (0.6) | -0.4 (0.9)
  Change from Baseline at Week 2: number analyzed (Participants) | 39 | 37 | 33 | 45
  Change from Baseline at Week 2 | -0.3 (0.8) | -0.3 (0.7) | -0.4 (0.6) | -0.9 (0.9)
  Change from Baseline at Week 4: number analyzed (Participants) | 39 | 35 | 30 | 40
  Change from Baseline at Week 4 | -0.1 (0.9) | -0.5 (0.8) | -0.6 (1.0) | -0.9 (0.9)
  Change from Baseline at Week 6: number analyzed (Participants) | 30 | 30 | 24 | 30
  Change from Baseline at Week 6 | -0.3 (0.8) | -0.5 (0.9) | -0.5 (1.1) | -0.9 (0.6)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Change from Baseline at Week 8 | -0.3 (0.8) | -0.5 (0.7) | -0.7 (0.9) | -0.7 (1.0)
  Change from Baseline at Week 14: number analyzed (Participants) | 12 | 18 | 13 | 17
  Change from Baseline at Week 14 | -0.3 (1.4) | -0.6 (0.7) | -1.0 (1.2) | -0.7 (1.0)
  Change from Baseline at Week 20: number analyzed (Participants) | 8 | 6 | 9 | 12
  Change from Baseline at Week 20 | -0.6 (0.7) | -0.3 (1.0) | -1.2 (1.1) | -0.9 (0.7)
  Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Change from Baseline at Week 26 | -0.8 (0.4) | 0.0 (0.0) | -1.0 (1.4) | -1.3 (0.8)
  Change from Baseline at Week 32: number analyzed (Participants) | 1 | 1 | 0 | 3
  Change from Baseline at Week 32 | -1.0 (NA) — The standard deviation was not evaluable for 1 participant. | -2.0 (NA) — The standard deviation was not evaluable for 1 participant. |  | -2.0 (1.0)
  Change from Baseline at End of the Study Visit (Week 43 or before) | -0.2 (1.1) | -0.6 (0.9) | -0.7 (1.1) | -0.9 (1.0)

3. Secondary Outcome: Mean Change From Baseline in Patient Global Impression - Severity of Depression Scale (PGI-S) Score
Description: The severity of illness was rated using a 7-point PGI-S. PGI-S scores range from 1 to 7, where 1=not depressed at all, 2=only occasionally depressed to a mild degree, 3=mildly depressed half the time, 4=moderately depressed most of the time, 5=moderately depressed almost all of the time, 6=severely depressed all the time, 7=extremely depressed all the time. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 14, 20, 26, 32 and End of the study visit (Week 43 or before)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 48
score on a scale
  Baseline | 2.8 (1.2) | 3.1 (1.2) | 3.3 (1.2) | 3.2 (1.4)
  Change from Baseline at Week 1: number analyzed (Participants) | 42 | 39 | 33 | 45
  Change from Baseline at Week 1 | 0.1 (0.8) | -0.2 (0.7) | -0.2 (0.8) | -0.6 (1.0)
  Change from Baseline at Week 2: number analyzed (Participants) | 39 | 37 | 33 | 45
  Change from Baseline at Week 2 | -0.2 (0.9) | -0.4 (0.9) | -0.4 (0.7) | -1.0 (1.2)
  Change from Baseline at Week 4: number analyzed (Participants) | 38 | 35 | 29 | 40
  Change from Baseline at Week 4 | 0.0 (1.1) | -0.5 (1.0) | -0.2 (1.0) | -0.9 (1.5)
  Change from Baseline at Week 6: number analyzed (Participants) | 30 | 29 | 23 | 30
  Change from Baseline at Week 6 | -0.1 (0.9) | -0.4 (1.3) | -0.4 (0.9) | -1.1 (1.1)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 17 | 26
  Change from Baseline at Week 8 | -0.2 (1.0) | -0.4 (1.0) | -0.3 (0.9) | -0.9 (1.5)
  Change from Baseline at Week 14: number analyzed (Participants) | 12 | 18 | 13 | 17
  Change from Baseline at Week 14 | -0.1 (1.8) | -0.2 (1.2) | -0.8 (1.2) | -0.9 (1.4)
  Change from Baseline at Week 20: number analyzed (Participants) | 8 | 6 | 9 | 12
  Change from Baseline at Week 20 | -0.4 (0.9) | -0.3 (1.2) | -1.0 (1.1) | -1.3 (1.3)
  Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Change from Baseline at Week 26 | 0.0 (1.4) | 0.0 (0.0) | -0.6 (2.1) | -1.0 (1.1)
  Change from Baseline at Week 32: number analyzed (Participants) | 1 | 1 | 0 | 3
  Change from Baseline at Week 32 | 0.0 (NA) — The standard deviation was not evaluable for 1 participant. | -1.0 (NA) — The standard deviation was not evaluable for 1 participant. |  | 0.0 (1.0)
  Change from Baseline at End of Study Visit (Week 43 or before) | -0.1 (1.2) | -0.3 (1.2) | -0.3 (1.2) | -0.9 (1.5)

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities: Heart rate [beats per minute (BPM)]: >120, increase >=15, <50, decrease >=15; systolic blood pressure [millimeter of mercury (mmHg)]: >180, increase >=20, <90, decrease >=20; diastolic blood pressure (mmHg): >105, increase >=15, <50, decrease >=15; orthostatic hypotension: >=20 mmHg decrease in systolic blood pressure and >=25 bpm increase in heart rate from supine to sitting; weight (kg) gain: increase >=7%; or weight loss: decrease >=7%. Only categories with at least 1 participant with event are reported.
Time Frame: Up to 40 weeks
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record. Number analyzed is the number of participants with at least one post-baseline numeric result for the given vital sign parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
Participants
  Orthostatic Hypotension (mmHg): number analyzed (Participants) | 44 | 41 | 36 | 48
  Orthostatic Hypotension (mmHg) | 0 | 0 | 1 | 0
  Weight (kg): Weight Gain >=7%: number analyzed (Participants) | 44 | 41 | 36 | 48
  Weight (kg): Weight Gain >=7% | 4 | 0 | 2 | 4
  Weight (kg): Weight Loss >=7%: number analyzed (Participants) | 44 | 41 | 36 | 48
  Weight (kg): Weight Loss >=7% | 5 | 2 | 1 | 2

5. Secondary Outcome: Mean Change From Baseline in Body Weight
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 14, 20, 26, 32 and End of the study visit (Week 43 or before)
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
kg
  Baseline | 93.0 (27.1) | 88.3 (23.5) | 87.0 (24.2) | 84.7 (22.6)
  Change from Baseline at Week 1: number analyzed (Participants) | 40 | 40 | 34 | 45
  Change from Baseline at Week 1 | 0.0 (2.4) | 0.1 (1.8) | 0.1 (1.2) | 0.1 (1.3)
  Change from Baseline at Week 2: number analyzed (Participants) | 39 | 36 | 32 | 40
  Change from Baseline at Week 2 | 0.5 (2.6) | 0.2 (2.1) | 0.2 (1.4) | 0.4 (1.5)
  Change from Baseline at Week 4: number analyzed (Participants) | 31 | 30 | 24 | 33
  Change from Baseline at Week 4 | 0.3 (3.8) | 0.4 (2.3) | 0.4 (1.4) | 0.2 (2.1)
  Change from Baseline at Week 6: number analyzed (Participants) | 26 | 26 | 19 | 25
  Change from Baseline at Week 6 | 0.3 (4.5) | 0.1 (2.9) | 0.3 (2.1) | 0.3 (2.8)
  Change from Baseline at Week 8: number analyzed (Participants) | 17 | 20 | 16 | 22
  Change from Baseline at Week 8 | -0.0 (5.5) | -0.5 (3.2) | 0.4 (2.7) | 0.2 (2.7)
  Change from Baseline at Week 14: number analyzed (Participants) | 9 | 8 | 9 | 13
  Change from Baseline at Week 14 | 2.0 (5.1) | -0.9 (4.8) | 0.7 (3.0) | 0.6 (4.3)
  Change from Baseline at Week 20: number analyzed (Participants) | 5 | 2 | 6 | 6
  Change from Baseline at Week 20 | 3.8 (2.6) | 2.0 (1.6) | 0.4 (5.7) | 1.4 (1.4)
  Change from Baseline at Week 26: number analyzed (Participants) | 1 | 1 | 0 | 3
  Change from Baseline at Week 26 | 5.7 (NA) — The standard deviation was not evaluable for 1 participant. | 1.4 (NA) — The standard deviation was not evaluable for 1 participant. |  | 3.3 (0.5)
  Change from Baseline at Week 32: number analyzed (Participants) | 0 | 1 | 0 | 0
  Change from Baseline at Week 32 |  | -3.6 (NA) — The standard deviation was not evaluable for 1 participant. |  |
  Change from Baseline at Last Visit (Week 43 or before): number analyzed (Participants) | 43 | 39 | 35 | 46
  Change from Baseline at Last Visit (Week 43 or before) | -0.2 (4.7) | 0.1 (3.1) | 0.1 (4.0) | 1.0 (3.7)

6. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI)
Description: BMI= weight(kg)/[height(m)^2].
Time Frame: Baseline, Week 26 and End of the study visit (Week 43 or before)
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record. Number analyzed is the number of participants with at least one observation at the given timepoint.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
kg/m^2
  Baseline | 33.4 (8.6) | 30.9 (8.1) | 31.1 (7.6) | 30.7 (7.4)
  Change from Baseline at Week 26: number analyzed (Participants) | 1 | 1 | 0 | 3
  Change from Baseline at Week 26 | 2.3 (NA) — The standard deviation was not evaluable for 1 participant. | 0.4 (NA) — The standard deviation was not evaluable for 1 participant. |  | 1.2 (0.2)
  Change from Baseline at Last Visit (Week 43 or before): number analyzed (Participants) | 33 | 34 | 27 | 38
  Change from Baseline at Last Visit (Week 43 or before) | 0.0 (2.5) | -0.1 (1.1) | -0.1 (1.5) | 0.4 (1.7)

7. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Test Abnormalities
Description: The laboratory values were one of the parameters to measure the safety and tolerability of individual participants. Participants with potentially clinically significant lab values in serum chemistry, hematology, urinalyses and prolactin tests that were identified based on pre-defined criteria were reported. Any value outside the normal range was flagged for the attention of the investigator who assessed whether or not a flagged value is of clinical significance. The categories with at least one participants with abnormal lab value as assessed by the Investigator are reported.
Time Frame: Up to 40 weeks
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record. Number analyzed is the total number of participants with at least one post-baseline numeric result for the given lab test.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
Participants
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN: number analyzed (Participants) | 43 | 38 | 34 | 48
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN | 0 | 1 | 0 | 0
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN: number analyzed (Participants) | 43 | 38 | 34 | 48
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN | 0 | 1 | 0 | 0
  Bilirubin, Total [mg/deciliter(dL)]: ≥2.0: number analyzed (Participants) | 43 | 38 | 34 | 48
  Bilirubin, Total [mg/deciliter(dL)]: ≥2.0 | 0 | 1 | 0 | 0
  Cholesterol, Total, Fasting (mg/dL): ≥240: number analyzed (Participants) | 39 | 34 | 29 | 44
  Cholesterol, Total, Fasting (mg/dL): ≥240 | 10 | 9 | 5 | 8
  Creatine phosphokinase (CPK), Total (U/L): ≥3 x ULN: number analyzed (Participants) | 43 | 38 | 34 | 48
  Creatine phosphokinase (CPK), Total (U/L): ≥3 x ULN | 0 | 1 | 0 | 1
  High-density Lipoprotein (HDL) Cholesterol, Fasting (mg/dL): ≤30: number analyzed (Participants) | 39 | 34 | 29 | 44
  High-density Lipoprotein (HDL) Cholesterol, Fasting (mg/dL): ≤30 | 0 | 0 | 2 | 1
  Low-density Lipoprotein (LDL) Cholesterol, Fasting (mg/dL): ≥160: number analyzed (Participants) | 38 | 35 | 28 | 44
  Low-density Lipoprotein (LDL) Cholesterol, Fasting (mg/dL): ≥160 | 6 | 5 | 4 | 8
  Triglycerides, Fasting (mg/dL): Men ≥160; Women ≥120: number analyzed (Participants) | 39 | 34 | 29 | 44
  Triglycerides, Fasting (mg/dL): Men ≥160; Women ≥120 | 24 | 16 | 14 | 25
  Urea Nitrogen (mg/dL); >= 30 mg/dL: number analyzed (Participants) | 43 | 38 | 34 | 48
  Urea Nitrogen (mg/dL); >= 30 mg/dL | 0 | 0 | 1 | 0
  Uric Acid (mg/dL): Men ≥10.5; Women ≥8.5: number analyzed (Participants) | 43 | 38 | 34 | 48
  Uric Acid (mg/dL): Men ≥10.5; Women ≥8.5 | 0 | 0 | 0 | 1
  Eosinophils (%): ≥10: number analyzed (Participants) | 43 | 37 | 33 | 48
  Eosinophils (%): ≥10 | 0 | 1 | 0 | 0
  Hematocrit (%): Female ≤32%; Male: ≤37% or 3 point decrease from baseline: number analyzed (Participants) | 43 | 36 | 32 | 44
  Hematocrit (%): Female ≤32%; Male: ≤37% or 3 point decrease from baseline | 0 | 1 | 1 | 0
  Hemoglobin (g/dL): Men ≤11.5; Women ≤9.5: number analyzed (Participants) | 43 | 37 | 33 | 48
  Hemoglobin (g/dL): Men ≤11.5; Women ≤9.5 | 1 | 0 | 1 | 0
  Prolactin [nanograms (ng)/mL]: >1 ULN: number analyzed (Participants) | 43 | 38 | 33 | 48
  Prolactin [nanograms (ng)/mL]: >1 ULN | 1 | 1 | 1 | 0

8. Secondary Outcome: Mean Change From Baseline in Laboratory Test Results: Prolactin
Description: Prolactin is a hormone released by the pituitary gland. The prolactin test measures the amount of prolactin in the blood. Prolactin is responsible for the breast growth and milk production during pregnancy and after birth. The normal prolactin levels range from 20 to 25 ng/mL in males and females and 80 to 400 ng/mL in pregnant women. A negative mean change from Baseline indicates reduction in the prolactin levels.
Time Frame: Baseline, Weeks 8, 26, and End of the study visit (Week 43 or before)
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record. Number analyzed is the total number of participants with at least one observation of the given parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
ng/mL
  Mean Change from Baseline at Week 8: number analyzed (Participants) | 17 | 20 | 16 | 21
  Mean Change from Baseline at Week 8 | 0.52 (3.94) | 0.31 (4.37) | 0.62 (3.26) | -1.10 (6.88)
  Mean Change from Baseline at Week 26: number analyzed (Participants) | 1 | 1 | 0 | 3
  Mean Change from Baseline at Week 26 | -0.79 (NA) — The standard deviation was not evaluable for 1 participant. | -2.75 (NA) — The standard deviation was not evaluable for 1 participant. |  | -0.75 (0.52)
  Mean Change from Baseline at Week Last Visit (Week 43 or before): number analyzed (Participants) | 43 | 38 | 33 | 46
  Mean Change from Baseline at Week Last Visit (Week 43 or before) | 0.37 (4.37) | 1.33 (4.71) | 0.30 (3.25) | -0.49 (5.57)

9. Secondary Outcome: Mean Change From Baseline in Laboratory Test Results: Hemoglobin A1c (HbA1c)
Description: The HbA1c is also known as glycosylated hemoglobin. It is the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound. The mean change in the value of HbA1c was analyzed relative to Baseline. The HbA1c of <6.0% signifies the normal blood glucose level. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline, Week 8, and End of the study visit (Week 43 or before)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 1 | 1 | 0 | 0
percentage of HbA1c
  Mean Change from Baseline at Week 8: number analyzed (Participants) | 0 | 1 | 0 | 0
  Mean Change from Baseline at Week 8 |  | 0.30 (NA) — The standard deviation was not evaluable for 1 participant. |  |
  Mean Change from Baseline at Last Visit (Week 43 or before) | -0.30 (NA) — The standard deviation was not evaluable for 1 participant. | 0.30 (NA) — The standard deviation was not evaluable for 1 participant. |  |

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Incidence of clinically relevant abnormal ECG values were reported as change from Baseline in heart rate (Tachycardia - ≥15 beats per minute (bpm), Bradycardia ≤15 bpm; Rhythm (Sinus tachycardia ≥15 bpm increase, Sinus bradycardia decrease of ≥15 bpm from Baseline); Presence of - supraventricular premature beat; ventricular premature beat; supraventricular tachycardia; ventricular tachycardia; atrial fibrillation and flutter. Conduction - Presence of primary, secondary or tertiary atrioventricular block, left bundle-branch block, right bundle-branch block, pre-excitation syndrome, other intraventricular conduction blocked QRS ≥0.12 second increase of ≥0.02 second. Acute, subacute or old Infarction, Presence of myocardial ischemia, symmetrical T-wave inversion. Increase in QTc - QTc ≥450 msec ≥10% increase. Any clinically significant change from Baseline assessed by the Investigator are reported. Only categories with at least 1 participant with event are reported.
Time Frame: Up to 40 weeks
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record. Number analyzed is the total number of participants with baseline and at least one post-baseline numeric result for the given ECG parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
Participants
  Bradycardia: Decrease of ≥15 bpm: number analyzed (Participants) | 42 | 37 | 34 | 46
  Bradycardia: Decrease of ≥15 bpm | 1 | 0 | 0 | 0
  Sinus Bradycardia: Decrease of ≥15 bpm: number analyzed (Participants) | 42 | 37 | 34 | 46
  Sinus Bradycardia: Decrease of ≥15 bpm | 1 | 0 | 0 | 0
  Supraventricular Premature Beat: Not Present to Present: number analyzed (Participants) | 42 | 37 | 34 | 46
  Supraventricular Premature Beat: Not Present to Present | 1 | 0 | 1 | 0
  Ventricular Premature Beat: Not Present to Present: number analyzed (Participants) | 42 | 37 | 34 | 46
  Ventricular Premature Beat: Not Present to Present | 0 | 1 | 1 | 0
  1° Atrioventricular Block: Increase of ≥0.05 second: number analyzed (Participants) | 42 | 37 | 34 | 46
  1° Atrioventricular Block: Increase of ≥0.05 second | 0 | 1 | 0 | 0
  Right Bundle-branch Block: Not Present to Present: number analyzed (Participants) | 42 | 37 | 34 | 46
  Right Bundle-branch Block: Not Present to Present | 1 | 0 | 0 | 1
  Myocardial Ischemia: Not Present to Present: number analyzed (Participants) | 42 | 37 | 34 | 46
  Myocardial Ischemia: Not Present to Present | 1 | 0 | 0 | 0
  Symmetrical T-wave Inversion: Not Present to Present: number analyzed (Participants) | 42 | 37 | 34 | 46
  Symmetrical T-wave Inversion: Not Present to Present | 3 | 1 | 0 | 0
  QTcB: number analyzed (Participants) | 42 | 37 | 34 | 46
  QTcB | 1 | 1 | 2 | 0
  QTcF: number analyzed (Participants) | 42 | 37 | 34 | 46
  QTcF | 0 | 1 | 2 | 1
  QTcN: number analyzed (Participants) | 42 | 37 | 34 | 46
  QTcN | 0 | 1 | 1 | 0

11. Secondary Outcome: Number of Participants With Potentially Clinically Significant Physical Examination Findings
Time Frame: Up to 40 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Mean Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS is a 12-item scale. The first 10 -items are rated from 0 to 4 (0=best, 4=worst). An item score of 0, depending on the item, either means: no abnormal involuntary movement (AIM), or no incapacitation due to AIM, or no awareness of AIM. An item score of 4 either means: severe AIM, or severe incapacitation due to AIM, or being aware of, and severe distress caused by AIM. Items 11 and 12, related to dental status, have dichotomous responses, 0=no and 1=yes. The AIMS Total Score is the sum of the ratings for the first seven items. The possible total scores are from 0 to 28, where a higher score indicates worst outcome. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 14, 20, 26, 32 and End of the study visit (Week 43 or before)
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record. Number analyzed is the number of participants with data available at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
score on a scale
  Baseline | 0.1 (0.5) | 0.0 (0.2) | 0.1 (0.3) | 0.1 (0.3)
  Change from Baseline at Week 4: number analyzed (Participants) | 39 | 35 | 30 | 40
  Change from Baseline at Week 4 | -0.1 (0.5) | -0.0 (0.2) | 0.0 (0.2) | 0.2 (1.1)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Change from Baseline at Week 8 | -0.1 (0.6) | 0.0 (0.0) | 0.0 (0.0) | -0.1 (0.4)
  Change from Baseline at Week 20: number analyzed (Participants) | 8 | 6 | 9 | 12
  Change from Baseline at Week 20 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | -0.2 (0.6)
  Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Change from Baseline at Week 26 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Change from Baseline at Week 32: number analyzed (Participants) | 1 | 1 | 0 | 3
  Change from Baseline at Week 32 | 0.0 (NA) — Standard deviation was not estimable for 1 participant. | 0.0 (NA) — Standard deviation was not estimable for 1 participant. |  | 0.0 (0.0)
  Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 44 | 39 | 35 | 48
  Change from Baseline at End of Study Visit (Week 43 or before) | -0.0 (0.5) | -0.0 (0.2) | -0.0 (0.4) | -0.0 (0.3)

13. Secondary Outcome: Mean Change From Baseline in Simpson-Angus Scale (SAS) Total Score
Description: The SAS is a rating scale used to measure extrapyramidal symptoms (EPS). The SAS is a 10-item scale, with each item rated from 1 to 5, with 1 being normal and 5 being the worst. The SAS total score is the sum of ratings for all 10 items, with possible total scores from 10 to 50. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 14, 20, 26, 32 and End of the study visit (Week 43 or before)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
score on a scale
  Baseline | 10.1 (0.3) | 10.0 (0.2) | 10.3 (0.7) | 10.1 (0.5)
  Change from Baseline at Week 4: number analyzed (Participants) | 39 | 35 | 30 | 40
  Change from Baseline at Week 4 | 0.0 (0.3) | 0.3 (0.7) | 0.0 (0.7) | 0.1 (0.5)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Change from Baseline at Week 8 | -0.1 (0.4) | 0.2 (0.5) | -0.1 (0.7) | -0.0 (1.0)
  Change from Baseline at Week 20: number analyzed (Participants) | 8 | 6 | 9 | 12
  Change from Baseline at Week 20 | 0.0 (0.0) | 0.0 (0.0) | -0.3 (0.7) | -0.3 (0.6)
  Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Change from Baseline at Week 26 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | -0.3 (0.8)
  Change from Baseline at Week 32: number analyzed (Participants) | 1 | 1 | 0 | 3
  Change from Baseline at Week 32 | 0.0 (NA) — The standard deviation was not evaluable for 1 participant. | 0.0 (NA) — The standard deviation was not evaluable for 1 participant. |  | -0.7 (1.2)
  Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 44 | 39 | 35 | 48
  Change from Baseline at End of Study Visit (Week 43 or before) | 0.1 (1.1) | 0.3 (0.8) | 0.1 (1.1) | -0.0 (0.5)

14. Secondary Outcome: Mean Change From Baseline in Barnes Akathisia Rating Scale (BARS) Global Clinical Assessment of Akathisia (Item 4) Score
Description: The BARS is used to assess the presence and severity of akathisia. This scale consists of 4 items. Only item 4, the 'Global Clinical Assessment of Akathisia', was evaluated for this outcome measure. This item is rated on a 6-point scale, with 0 being best (absent) and 5 being worst (severe akathisia). A negative mean change from Baseline indicates improvement.
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 14, 20, 26, 32 and End of the study visit (Week 43 or before)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
score on a scale
  Baseline | 0.2 (0.5) | 0.1 (0.4) | 0.4 (0.8) | 0.1 (0.4)
  Change from Baseline at Week 4: number analyzed (Participants) | 39 | 35 | 30 | 39
  Change from Baseline at Week 4 | 0.1 (0.6) | 0.3 (0.7) | 0.0 (0.8) | 0.2 (0.6)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Change from Baseline at Week 8 | -0.1 (0.6) | 0.3 (1.0) | -0.1 (1.1) | -0.0 (0.6)
  Change from Baseline at Week 20: number analyzed (Participants) | 8 | 6 | 9 | 12
  Change from Baseline at Week 20 | -0.1 (0.4) | -0.2 (0.4) | -0.4 (1.0) | -0.3 (0.9)
  Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Change from Baseline at Week 26 | -0.2 (0.4) | -0.5 (0.7) | 0.0 (0.0) | 0.0 (0.0)
  Change from Baseline at Week 32: number analyzed (Participants) | 1 | 1 | 0 | 3
  Change from Baseline at Week 32 | 0.0 (NA) — The standard deviation was not evaluable for 1 participant. | -1.0 (NA) — The standard deviation was not evaluable for 1 participant. |  | -0.3 (0.6)
  Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 44 | 39 | 35 | 47
  Change from Baseline at End of Study Visit (Week 43 or before) | -0.0 (0.6) | 0.3 (0.9) | -0.1 (1.1) | 0.0 (0.5)

15. Secondary Outcome: Percentage of Participants With Suicidal Ideation in Each Item as Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The suicidal ideation compared to Baseline was measured by an increase in suicidal ideation category (1-5 on the C-SSRS) during treatment from the maximum suicidal ideation category at Baseline, or any suicidal ideation during treatment if there is none at Baseline. C-SSRS is used to assess whether participant experienced suicidal ideation (Question 1: wish to be dead; Question 2: non-specific active suicidal thoughts; Question 3: active suicidal ideation with any methods (not plan) without intent to act; Question 4: active suicidal ideation with some intent to act, without specific plan; Question 5: active suicidal ideation with specific plan and intent). A negative change from Baseline indicates improvement. Only those categories and timepoints which have data are reported.
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 14 and Last Visit (Week 43 or before)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
percentage of participants
  Question 1: Baseline | 0.0 | 12.2 | 8.3 | 4.1
  Question 1: Week 1 | 0.0 | 2.4 | 2.8 | 0.0
  Question 1: Week 2 | 0.0 | 2.4 | 2.8 | 0.0
  Question 1: Week 4 | 2.3 | 4.9 | 2.8 | 0.0
  Question 1: Week 6 | 2.3 | 4.9 | 2.8 | 0.0
  Question 1: Week 8 | 0.0 | 0.0 | 2.8 | 2.0
  Question 1: Week 14 | 2.3 | 0.0 | 0.0 | 0.0
  Question 1: Last Visit (Week 43 or before) | 2.3 | 2.4 | 5.6 | 0.0
  Question 2: Week 8 | 0.0 | 0.0 | 0.0 | 2.0
  Question 2: Week 14 | 2.3 | 0.0 | 0.0 | 0.0
  Question 2: Last Visit (Week 43 or before) | 0.0 | 0.0 | 2.8 | 0.0
  Question 3: Week 14 | 2.3 | 0.0 | 0.0 | 0.0
  Question 3: Last Visit (Week 43 or before) | 0.0 | 0.0 | 2.8 | 0.0

16. Secondary Outcome: Mean Change From Baseline in Each Item as Measured by Massachusetts General Hospital Sexual Functioning Inventory (MGH SFI) Subscale Score
Description: The MGH SFI is a measure of a participant's self-reported sexual functioning. The MGH SFI included 5 questions at the baseline assessment, each addressing experiences over the last month: Question a) interest in sex, Question b) ability to get sexually aroused, Question c) ability to achieve orgasm, Question d) ability to get and maintain an erection, and Question e) overall sexual satisfaction. The MGH SFI at post-baseline visits included one additional question: Question f) overall improvement since the last medication change. Each question/item is rated from 1 through 6. For questions a) through e), a score of 1 indicates 'greater than normal', and 6 'totally absent'. For question f), a score of 1 indicates 'very much improved', and 6 'much worse'. All question scores are analyzed separately. No total or mean score is derived. Each subscale score ranges from 0 to 6, higher scores indicates worsening. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 8, 26 and End of the study visit (Week 43 or before)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 44 | 41 | 36 | 49
score on a scale
  Question a: Baseline | 4.2 (1.7) | 3.8 (1.5) | 4.4 (1.4) | 3.6 (1.6)
  Question a: Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Question a: Change from Baseline at Week 8 | -0.1 (1.3) | -0.4 (0.9) | -0.4 (0.8) | -0.3 (1.1)
  Question a: Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Question a: Change from Baseline at Week 26 | -0.2 (0.4) | 0.0 (0.0) | -0.4 (1.1) | 0.0 (0.0)
  Question a: Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 43 | 38 | 35 | 47
  Question a: Change from Baseline at End of Study Visit (Week 43 or before) | -0.1 (1.1) | -0.3 (1.1) | -0.4 (1.2) | -0.4 (1.2)
  Question b: Baseline | 3.9 (1.7) | 3.7 (1.5) | 4.1 (1.4) | 3.5 (1.6)
  Question b: Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Question b: Change from Baseline at Week 8 | 0.0 (0.9) | -0.2 (0.9) | -0.1 (0.9) | -0.3 (0.9)
  Question b: Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Question b: Change from Baseline at Week 26 | 0.2 (0.4) | 0.0 (0.0) | 0.0 (1.2) | -0.2 (0.4)
  Question b: Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 43 | 38 | 35 | 47
  Question b: Change from Baseline at End of Study Visit (Week 43 or before) | 0.1 (0.8) | -0.3 (1.0) | -0.2 (1.0) | -0.3 (1.1)
  Question c: Baseline | 4.0 (1.7) | 3.8 (1.5) | 4.1 (1.5) | 3.5 (1.6)
  Question c: Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Question c: Change from Baseline at Week 8 | -0.1 (1.0) | -0.3 (1.1) | -0.1 (0.9) | -0.2 (0.9)
  Question c: Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Question c: Change from Baseline at Week 26 | -0.2 (1.1) | 0.0 (0.0) | -0.2 (1.3) | -0.2 (0.4)
  Question c: Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 43 | 38 | 35 | 47
  Question c: Change from Baseline at End of Study Visit (Week 43 or before) | -0.0 (1.0) | -0.4 (1.1) | 0.0 (1.1) | -0.1 (1.1)
  Question d: Baseline: number analyzed (Participants) | 11 | 16 | 11 | 17
  Question d: Baseline | 2.5 (1.2) | 3.0 (1.4) | 3.6 (1.3) | 2.9 (1.3)
  Question d: Change from Baseline at Week 8: number analyzed (Participants) | 6 | 8 | 5 | 10
  Question d: Change from Baseline at Week 8 | 0.0 (0.0) | 0.0 (0.5) | -0.4 (0.5) | -0.2 (0.4)
  Question d: Change from Baseline at Week 26: number analyzed (Participants) | 1 | 2 | 1 | 2
  Question d: Change from Baseline at Week 26 | 0.0 (NA) — The standard deviation was not evaluable for 1 participant. | 0.5 (0.7) | 0.0 (NA) — The standard deviation was not evaluable for 1 participant. | 0.0 (0.0)
  Question d: Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 10 | 15 | 9 | 16
  Question d: Change from Baseline at End of Study Visit (Week 43 or before) | 0.1 (0.3) | 0.0 (0.5) | 0.1 (0.9) | -0.1 (0.8)
  Question e: Baseline | 4.2 (1.7) | 3.9 (1.6) | 4.4 (1.3) | 3.7 (1.6)
  Question e: Change from Baseline at Week 8: number analyzed (Participants) | 26 | 23 | 18 | 26
  Question e: Change from Baseline at Week 8 | -0.1 (1.1) | -0.3 (0.8) | -0.3 (0.8) | -0.2 (1.1)
  Question e: Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Question e: Change from Baseline at Week 26 | -0.4 (0.5) | 0.5 (0.7) | -0.4 (1.1) | 0.0 (0.6)
  Question e: Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 43 | 38 | 34 | 47
  Question e: Change from Baseline at End of Study Visit (Week 43 or before) | -0.1 (0.9) | -0.3 (1.2) | -0.3 (1.4) | -0.3 (1.4)
  Question f: Baseline | 3.3 (0.9) | 3.5 (1.2) | 3.4 (1.1) | 3.6 (1.2)
  Question f: Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Question f: Change from Baseline at Week 8 | 0.1 (1.1) | -0.3 (1.1) | 0.2 (1.1) | -0.7 (1.7)
  Question f: Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Question f: Change from Baseline at Week 26 | -1.0 (0.7) | 0.0 (0.0) | 0.4 (1.9) | -0.8 (1.3)
  Question f: Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 43 | 38 | 34 | 47
  Question f: Change from Baseline at End of Study Visit (Week 43 or before) | -0.0 (1.0) | -0.2 (1.1) | -0.0 (1.6) | -0.6 (1.5)

17. Secondary Outcome: Mean Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) Overall General Subscore
Description: The Q-LES-Q-SF is a self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning with the help of 14 items of total 16 items of the scale. The overall general subscore is obtained using 14 items of the scale. Each item is scored on a 5-point scale, with 1= Very Poor; 2=Poor; 3=Fair; 4=Good; 5=Very Good. The raw scores are computed to an overall general subscore of 0 to 100 where lower scores indicate less enjoyment or satisfaction with the activity. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Week 8, 26 and End of the study visit (Week 43 or before)
Population: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record, with data available for analysis. Number analyzed is the number of participants with data available at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 43 | 41 | 36 | 49
score on a scale
  Baseline | 49.4 (14.7) | 50.2 (19.9) | 47.9 (16.8) | 52.2 (14.6)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 25
  Change from Baseline at Week 8 | 0.8 (10.4) | 3.6 (11.0) | 6.2 (9.9) | 9.5 (13.6)
  Change from Baseline at Week 26: number analyzed (Participants) | 4 | 2 | 5 | 6
  Change from Baseline at Week 26 | 0.8 (19.6) | -0.5 (2.1) | 6.2 (22.4) | 4.3 (17.7)
  Change from Baseline at End of Study visit (Week 43 or before): number analyzed (Participants) | 42 | 37 | 35 | 47
  Change from Baseline at End of Study visit (Week 43 or before) | 1.0 (14.1) | 5.0 (15.4) | 4.6 (14.3) | 10.0 (16.5)

18. Secondary Outcome: Mean Change From Baseline in Sheehan Disability Scale (SDS) Mean Total Score
Description: The SDS is a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores range from 0 through 10. The number most representative of how much each area was disrupted by symptoms was marked along the line from 0= not at all, to 10= extremely. For the work/school item, no response was to be entered if the participant did not work or go to school for reasons unrelated to the disorder and a response therefore not being applicable. The SDS Mean Score of 0 to 10 was calculated as an average of the three item scores. All three item scores needed to be available with the exception of the work/school item score when this item was not applicable. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 8, 26 and End of the study visit (Week 43 or before)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 43 | 41 | 36 | 49
score on a scale
  Baseline | 4.6 (2.6) | 4.3 (2.7) | 5.1 (2.7) | 3.8 (2.1)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 26
  Change from Baseline at Week 8 | -1.1 (2.1) | -0.8 (1.6) | -2.0 (2.4) | -1.4 (1.8)
  Change from Baseline at Week 26: number analyzed (Participants) | 5 | 2 | 5 | 6
  Change from Baseline at Week 26 | -1.9 (1.6) | 1.7 (2.4) | -2.6 (2.7) | -0.7 (4.6)
  Change from Baseline at End of Study visit (Week 43 or before): number analyzed (Participants) | 42 | 38 | 35 | 48
  Change from Baseline at End of Study visit (Week 43 or before) | -0.6 (2.1) | -0.5 (2.5) | -1.6 (2.8) | -1.6 (2.2)

19. Secondary Outcome: Mean Change From Baseline in Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) Total Score
Description: The CPFQ is a brief self-rated scale developed to measure cognitive and executive dysfunction in mood and anxiety disorders. It consists of 7 items. The CPFQ total score ranges from 7 to 42, with higher score representing less satisfaction in cognitive and physical functioning. A negative mean change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 8, 26 and End of the study visit (Week 43 or before)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
Number analyzed (Participants) | 43 | 41 | 34 | 49
score on a scale
  Baseline | 23.0 (6.1) | 22.1 (6.5) | 24.4 (5.3) | 22.0 (6.1)
  Change from Baseline at Week 8: number analyzed (Participants) | 26 | 24 | 18 | 25
  Change from Baseline at Week 8 | -1.3 (4.1) | -1.8 (2.6) | -2.2 (3.3) | -4.8 (7.7)
  Change from Baseline at Week 26: number analyzed (Participants) | 4 | 2 | 5 | 6
  Change from Baseline at Week 26 | -3.8 (3.5) | 2.0 (0.0) | -2.2 (5.6) | -2.5 (6.0)
  Change from Baseline at End of Study Visit (Week 43 or before): number analyzed (Participants) | 42 | 37 | 33 | 47
  Change from Baseline at End of Study Visit (Week 43 or before) | -1.0 (4.6) | -0.2 (4.8) | -2.6 (5.0) | -3.5 (7.6)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days post last dose (Up to 40 weeks)
Description: Safety Sample included all participants who received in the Treatment Phase at least one dose of aripiprazole/escitalopram combination medication as indicated on the dosing record.
Arm/Group | Prior Aripiprazole/Escitalopram Combination Therapy | Prior Escitalopram | Prior Aripiprazole | Prior Single-blind Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/41 | 0/36 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/44 | 4/41 | 0/36 | 0/49
Other Adverse Events (participants affected / at risk) | 18/44 | 27/41 | 33/36 | 31/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Aripiprazole/Escitalopram Combination Therapy (N=44) | Prior Escitalopram (N=41) | Prior Aripiprazole (N=36) | Prior Single-blind Escitalopram (N=49)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Aripiprazole/Escitalopram Combination Therapy (N=44) | Prior Escitalopram (N=41) | Prior Aripiprazole (N=36) | Prior Single-blind Escitalopram (N=49)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 7 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 4 | 4
Blood glucose increased (Investigations) | 0 | 3 | 0 | 0
Weight increased (Investigations) | 2 | 1 | 3 | 2
Akathisia (Nervous system disorders) | 2 | 4 | 3 | 6
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 2
Headache (Nervous system disorders) | 1 | 2 | 2 | 5
Sedation (Nervous system disorders) | 1 | 2 | 0 | 5
Somnolence (Nervous system disorders) | 4 | 2 | 3 | 2
Anxiety (Psychiatric disorders) | 1 | 3 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 3 | 1 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early due to Sponsor decision; no safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.